CLINICAL TRIAL: NCT05394532
Title: Effect of Steno Diabetes Dialogue Cards Teaching Instrument on Diabetes in Group Education on Blood Sugar Control in Adolescents With Type 1 Diabetes
Brief Title: Steno Diabetes Dialogue Cards Teaching on Group Education on Blood Sugar Control in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Lin, I-Hsiang, Master, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IHLin
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Type 1 Diabetes; HbA1c; Self-management
Keywords: type 1 diabetes mellitus; Steno Balance Card; group health education; blood sugar control; self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steno Diabetes Dialogue Cards (Experimental)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Common Education

SUMMARY:
The Type 1 diabetes is the autoimmunity system produces the antibody which starts to attack the B lymphocytes while the autoimmunity is also been attacked. When the autoimmunity system has been destoyed, the insulin couldn't be secreted normally. thus, the hyperglycaemia is caused. Then, the patients need to rely on the insulin injection throughout the lifetime. The main symptoms are the three mores （eat more, drink more and urinate more）, weight loss, urine sugar, lethargy, ketone bodies and ect. The most serious complications of the diabetes type 1 is the Diabetic ketoacidosis, DKA. It is caused by the severe infection or poor Glycemic Control. If the DKA happened, the patients need to be rescued in the ICU. is because it sometimes endager life. The diabetes type 1 patients rely on the insulin injection throughout the lifetime and a good habbit of diet, boold sugar controlling and exercise. The DKA happens when the boold sugar is not well controlled.

ELIGIBILITY:
Inclusion Criteria:

* 10-18years ord Type 1 DM.
* Able to read and write Chinese.

Exclusion Criteria:

* Communication and cognitive impairments.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  The subjects were 83 adolescents diagnosed with type 1 diabetes mellitus. The experiment group intervened with the Steno Balance Card method was better than the control group which received only general health education in terms of blood sugar control after 3 months .

SECONDARY OUTCOMES:
self management | 3 months
  There was in scores between the experimental and the control groups three months after intervention which means both health education methods improved the level of self-management in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fangyi Lin, Taipei, Beitou, Taiwan